CLINICAL TRIAL: NCT04726904
Title: Best Surgical Technique for Optimal Lead Placement in Sacral Neuromodulation - a Comparative Cadaver Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christopher Dawoud, Dr.med.univ., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2219/2018
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Faecal Incontinence
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional lead placement (Other): The cadaver is placed in the prone position. The exact location for insertion of the needle is defined with the conventional technique.
  Interventions: Procedure: Sacral neuromodulation in conventional implantation technique

INTERVENTIONS:
Procedure: Sacral neuromodulation in conventional implantation technique — Sacral neuromodulation is implanted with the patients in a prone position, then the insert point of the needle is decided according to anatomical landmarks; afterwards, the lead will be inserted.

SUMMARY:
Sacral neuromodulation (SNM) is an established treatment option for patients with faecal incontinence. The location of the stimulating electrode is considered to be essential for treatment success. The purpose of this study was to evaluate the position of SNM electrodes after using the conventional implantation technique and to compare our results with those of the preliminary study, where the standardised fluoroscopy-guided implantation technique was used.

In this cadaver study, SNM electrodes will be implanted bilaterally in 5 lower body specimens. After electrode placement the pelvis was dissected to describe the exact position of the SNM electrodes.

DETAILED DESCRIPTION:
Sacral neuromodulation (SNM) is an established treatment option for patients with faecal incontinence. The location of the stimulating electrode is considered to be essential for treatment success. The purpose of this study was to evaluate the position of SNM electrodes after using the conventional implantation technique and to compare our results with those of the preliminary study, where the standardised fluoroscopy-guided implantation technique was used.

However, to date no studies exist comparing different surgical techniques. The present cadaver study was designed to assess the distance between lead and sacral nerves by comparing two different surgical techniques: the new fluoroscopy guided "H" technique and the commonly conducted non radiological lead implantation using anatomical landmarks.

In this cadaver study, SNM electrodes will be implanted bilaterally in 5 lower body specimens.Afterwards the cadaver will be dissected and the exact location to the nerve, as well as a perforation of the sacral fascia will be noted.

The results will be compared to the preliminary study of Mueller et al., where they used the new fluoroscopy guided "H" technique in five cadavers.

ELIGIBILITY:
Inclusion Criteria:

* Cadaver study
* All of these individuals had donated their bodies to medical education and research in form of an informed consent.

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Distance lead to nerve | 1 week
  The exact distance (mm) will be assessed from the lead to the nerve

SECONDARY OUTCOMES:
Neuroforamen | 1 week
  The inserted neuroforamen will be assessed.
Sacral fascia | 1 week
  A perforation throw the sacral fascia will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dawoud, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Muller C, Reissig LF, Argeny S, Weninger WJ, Riss S. Standardized fluoroscopy-guided implantation technique enables optimal electrode placement in sacral neuromodulation: a cadaver study. Tech Coloproctol. 2021 Feb;25(2):215-221. doi: 10.1007/s10151-020-02364-w. Epub 2020 Nov 19. PMID 33211205